CLINICAL TRIAL: NCT01407003
Title: A Randomized, Double-blind, Placebo-controlled, 4-part, Interwoven Single- and Multiple-ascending Dose Study to Assess Safety, Tolerability, PK and PD of LIK066 in Healthy Subjects and in Patients With T2DM
Brief Title: Safety, Tolerability, Pharmacokinetics (PK) and Pharmacodynamics (PD) Assessment of LIK066 in Healthy Subjects and in Patients With Type 2 Diabetes Mellitus (T2DM)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: CLIK066X2101
Record Dates: First submitted 2011-07-20; First posted 2011-08-01 (Estimated); Last update posted 2020-12-19 (Actual); Status verified 2014-04

CONDITIONS: Type 2 Diabetes Mellitus (T2DM)
Keywords: T2DM, blood glucose, OGTT, LIK066
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — licogliflozin

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (4):
- LIK066 in healthy subjects (Experimental)
  Interventions: Drug: LIK066
- Matching placebo in healthy subjects (Placebo Comparator)
  Interventions: Drug: Placebo
- LIK066 in patients with type 2 diabetes mellitus (Experimental)
  Interventions: Drug: LIK066
- Matching placebo in patients with type 2 diabetes mellitus (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: LIK066 — Participants will receive a single or multiple doses of LIK066
  Arms: LIK066 in healthy subjects; LIK066 in patients with type 2 diabetes mellitus
Drug: Placebo — Participants will receive a single or multiple doses of a matching placebo
  Arms: Matching placebo in healthy subjects; Matching placebo in patients with type 2 diabetes mellitus

SUMMARY:
This study will assess safety, tolerability, and effect of LIK066 on blood glucose in healthy subjects and in patients with T2DM.

ELIGIBILITY:
Inclusion Criteria:

* Parts I and III: Healthy male and female subjects age 18 to 55 years of age included, and in good health as determined by past medical history, physical examination, electrocardiogram, and laboratory tests at screening.
* Parts II and IV: Patients, age 18-65 years, must have been diagnosed with T2DM at least 8 weeks prior to screening with HbA1c 6.5 to 10.0%, inclusive, at screening.
* Fasting plasma glucose ≤250mg/dL at screening and baseline.
* If treated with metformin, patients must be on a stable dose for 12 weeks prior to randomization and maintain the dose until the end of the study.

Exclusion Criteria; all parts:

* Patients with type 1 diabetes mellitus.
* Patients with history of acute diabetic complications within the 6 months prior to screening.
* Women of child-bearing potential.
* Patients with signs or symptoms of significant diabetic complications.
* Patients treated with certain blood pressure or lipid lowering medications unless patients have been on stable doses for the 12 weeks prior to dosing.
* History of drug or alcohol abuse within the 12 months prior to dosing.
* Any surgical or medical condition, acute or unstable chronic disease which may, based on the investigator's opinion, jeopardize the patient in case of participation in the study.

Other protocol-defined inclusion/exclusion criteria may apply

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 138 (Actual)
Dates: Start 2011-06; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of single and multiple dose(s) of LIK066: number of patients with adverse events and changes from baseline in vital signs, ECG and clinical labs (blood chemistry, hematology and urinalysis). | Daily during treatment

SECONDARY OUTCOMES:
Change in fasting and post-challenge plasma glucose after 2 weeks of treatment | Baseline and End of Treatment
Pharmacokinetics: to measure the study drug concentration in blood and urine samples to be collected after drug administration | Day 1 and End of Treatment
Change in fasting and post-challenge plasma glucose after a single dose and 2 weeks of treatment | Baseline and End of Treatment

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (1):
- Novartis Investigative Site, Miami, Florida, United States

REFERENCES:
- See also: Results for CLIK066X2101 from the Novartis Clinical Trials website — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=11104